CLINICAL TRIAL: NCT07097948
Title: Toripalimab Combined With Chemotherapy as Adjuvant Therapy for Incidental Small Cell Lung Cancer After Radical Resection of Lung Cancer: A Single-Center, Randomized Controlled Clinical Study
Brief Title: Toripalimab Combined With Chemotherapy as Adjuvant Therapy for Incidental Small Cell Lung Cancer After Radical Resection of Lung Cancer: A Single-Center, Randomized Controlled Clinical Study Protocol Number: LungMate-033
Acronym: Adjuvant
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-033
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Incidental Small Cell Lung Cancer; Toripalimab Adjuvant Therapy Evaluation
Keywords: Small cell lung cancer; Postoperative adjuvant therapy; Toripalimab; Immunological maintenance; Recurrence
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — Etoposide; Platinum; toripalimab

STUDY DESIGN:
Intervention Model Description: For patients with postoperatively incidentally detected small cell lung cancer, all enrolled patients will be randomized into two groups: one group receiving toripalimab combined with platinum-based chemotherapy, and the other group receiving platinum-based chemotherapy alone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative Adjuvant Chemotherapy (Active Comparator): In this arm, enrolled subjects will receive postoperative adjuvant chemotherapy, totaling 4 cycles, with each cycle lasting 3 weeks.
  Interventions: Drug: Etoposide; Drug: Platinum
- Postoperative Chemotherapy Combined with Toripalimab Maintenance (Experimental): In this arm, enrolled subjects will first receive postoperative chemotherapy (4 cycles, 3 weeks per cycle), followed by toripalimab for immunological maintenance therapy, administered once every 3 weeks.
  Interventions: Drug: Etoposide; Drug: Platinum; Drug: Toripalimab

INTERVENTIONS:
Drug: Etoposide — Specified dose on specified days.
Drug: Platinum — Specified dose on specified days.
Drug: Toripalimab — Specified dose on specified days.
  Arms: Postoperative Chemotherapy Combined with Toripalimab Maintenance

SUMMARY:
Small cell lung cancer (SCLC) is highly malignant and aggressive, with most patients presenting with metastases at diagnosis. For postoperatively incidentally detected SCLC (identified unexpectedly in pathological examinations after surgery), conventional adjuvant chemoradiotherapy has shown limited efficacy, characterized by high recurrence rates and suboptimal long-term survival.Notably, advances in immunotherapy have transformed SCLC management. The EXTENTORCH trial, a pivotal study published in JAMA Oncology, demonstrated that toripalimab plus chemotherapy significantly improved outcomes in extensive-stage SCLC (ES-SCLC), achieving a reduced risk of progression or death (HR=0.67, 95% CI 0.54-0.82, P<0.001) with manageable safety, marking a substantial therapeutic breakthrough. Given the proven efficacy of toripalimab in ES-SCLC, there is a strong rationale to extend this strategy to postoperatively incidentally detected SCLC. This trial aims to evaluate the efficacy and safety of toripalimab as adjuvant maintenance therapy in this cohort, with the objective of reducing recurrence and enhancing long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form;
2. Aged ≥ 18 years;
3. Patients with definitely incidental SCLC confirmed by pathological results after radical resection of lung cancer;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Life expectancy is at least 12 weeks;
6. Good function of other major organs (liver, kidney, hematological system, etc.);
7. Fertile female patients must undergo a pregnancy test within 7 days before the start of treatment with a negative result; and reliable contraceptive measures (such as intrauterine devices, contraceptives and condoms) should be used during the trial and within 30 days after its completion;
8. Fertile male subjects must use condoms for contraception during the trial and within 30 days after its completion.

Exclusion Criteria:

1. Patients with a malignancy other than SCLC within five years prior to the start of this trial;
2. Participants with any unstable systemic disease (including uncontrolled hypertension, severe arrhythmia, etc.);
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with active hepatitis B, hepatitis C or HIV;
6. Participants with Interstitial lung disease currently;
7. Pregnant or lactating women;
8. Any malabsorption;
9. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | up to 60 months
  Defined as the time from the initiation of treatment to the first confirmed disease recurrence or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 60 months
  Defined as the time from the date of initial treatment to death from any cause. For patients still alive at the time of analysis, the date of last contact will be used as the censoring date. Survival curves will be estimated using the Kaplan-Meier method.
Health related quality of life (HRQol)：EORTC-QLQ-C30 | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 , Version 3). EORTC's QLQ-C30 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options.
Health related quality of life (HRQol)：LC13 | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (LC13, Version 3).The items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.